CLINICAL TRIAL: NCT03385447
Title: The Physiological and Cognitive Effects of Faculty/Staff Exercise Program in a University Setting
Brief Title: The Effects of Faculty/Staff Exercise Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kent State University (Other)
Responsible Party: Principal Investigator, Duane Corbett, Graduate Assistant, Kent State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 13-329
Record Dates: First submitted 2017-12-04; First posted 2017-12-28 (Actual); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Cardiovascular Risk Factor; Sedentary Lifestyle; Physical Activity
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical Activity (Experimental): Participants were subjected to a 12-week exercise program targeting the federal physical activity guidelines.
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — Participants underwent 12-weeks of exercise prescription aimed at the federal guidelines (3 days/week).

SUMMARY:
This study focuses on analyzing the data collected from participants in the Faculty/Staff Exercise Program to determine the success and quantifying the results of the program. The investigators are interested in the effectiveness of this program on multiple levels, individual and group, as it is the first of its kind - an exercise program targeting the faculty and staff at a university.

DETAILED DESCRIPTION:
This study focuses on analyzing the data collected from participants in the Faculty/Staff Exercise Program to determine the success and quantifying the results of the program. The investigators are interested in the effectiveness of this program on multiple levels, individual and group, as it is the first of its kind - an exercise program targeting the faculty and staff at a university. Participants were regular attendees in either a 6am or 12pm exercise program session. Data included both measures of physical health as well as cognitive health. Measures of physical health included the assessment of body fat using the skin-fold method of analysis (3-site). Cholesterol was measured via blood draw analysis. This was done at the Kent State University Exercise Physiology Laboratory by certified research staff. A 6 minute walk test was completed to measure aerobic capacity. Flexibility was assessed via the sit-and-reach test while anaerobic strength and endurance were assessed using sit-up and curl-up tests. Assessment of balance was done using a Biodex Balance System.

Assessments of cognitive health included several questionnaires that asked questions related to sleep habits, stress levels, and mood. In addition, each participant was given a MOVband to track physical activity. The device was worn during waking hours for all days of participation.The data from the MOVband was auto-uploaded to a computer program for tracking so that no manual entry was necessary.

ELIGIBILITY:
Inclusion Criteria:

* age 21-65 years
* current faculty/staff member
* no contraindications to exercise
* sedentary prior to enrollment

Exclusion Criteria:

* age <21 years, >65 years
* non faculty/staff member
* contraindications to exercise
* regular exercise participation prior to enrollment

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-06-26 (Actual); Primary Completion 2013-10-11 (Actual); Study Completion 2013-10-11 (Actual)

PRIMARY OUTCOMES:
Height | Assessed once at baseline.
  Objectively measured height in meters using a standard clinical stadiometer.
Weight | Change from baseline weight at 4-weeks, 8-weeks, and 12-weeks follow-up.
  Objectively measured weight in kilograms using a standard clinical scale.
Systolic Blood Pressure | Change from baseline systolic blood pressure at 4-weeks, 8-weeks, and 12-weeks follow-up.
  Objectively measured systolic blood pressure in millimeters of Mercury using a standard Mercury sphygmomanometer.
Diastolic Blood Pressure | Change from baseline diastolic blood pressure at 4-weeks, 8-weeks, and 12-weeks follow-up.
  Objectively measured diastolic blood pressure in millimeters of Mercury using a standard Mercury sphygmomanometer.
High-Density Lipoprotein | Change from baseline high-density lipoprotein at 4-weeks, 8-weeks, and 12-weeks follow-up.
  Objectively measured high-density lipoprotein in milligrams per deciliter using a standard assay kit.
Low-Density Lipoprotein | Change from baseline low-density lipoprotein at 4-weeks, 8-weeks, and 12-weeks follow-up.
  Objectively measured low-density lipoprotein in milligrams per deciliter using a standard assay kit.
Total Serum Cholesteral | Change from baseline total serum cholesterol at 4-weeks, 8-weeks, and 12-weeks follow-up.
  Objectively measured total serum cholesterol in milligrams per deciliter using a standard assay kit.
Impaired Fasting Glucose | Change from baseline impaired fasting glucose at 4-weeks, 8-weeks, and 12-weeks follow-up.
  Objectively measured impaired fasting glucose in milligrams per deciliter using a standard assay kit.

SECONDARY OUTCOMES:
Accelerometer-Based Physical Activity | Change from baseline accelerometer-based physical activity 4-weeks, 8-weeks, and 12-weeks follow-up using 1-minute epochs.
  Assessment of accelerometer-based physical activity outcome measures (e.g., steps per day).

OTHER OUTCOMES:
Sleep Quality (Pittsburgh Sleep Quality Index) | Change from baseline sleep quality at 4-weeks, 8-weeks, and 12-weeks follow-up.
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval.
Depression (Depression, Anxiety, and Stress Scale-21) | Change from baseline depression at 4-weeks, 8-weeks, and 12-weeks follow-up.
  The depression, anxiety, and stress scale-21 (DASS-21) is a clinical assessment that measures the three related states of depression, anxiety and stress.
Anxiety (Depression, Anxiety, and Stress Scale-21) | Change from baseline anxiety at 4-weeks, 8-weeks, and 12-weeks follow-up.
  The depression, anxiety, and stress scale-21 (DASS-21) is a clinical assessment that measures the three related states of depression, anxiety and stress.
Stress (Depression, Anxiety, and Stress Scale-21) | Change from baseline stress at 4-weeks, 8-weeks, and 12-weeks follow-up.
  The depression, anxiety, and stress scale-21 (DASS-21) is a clinical assessment that measures the three related states of depression, anxiety and stress.
Mood (Profile of Mood States) | Change from baseline mood at 4-weeks, 8-weeks, and 12-weeks follow-up.
  The Profile of Mood States (POMS) is a psychological rating scale used to assess transient, distinct mood states.
Quality of Life (36-Item Short Form Survey) | Change from baseline quality of life at 4-weeks, 8-weeks, and 12-weeks follow-up.
  The 36-item short form survey (SF-36) is a set of generic, coherent, and easily administered quality-of-life measures.

CONTACTS AND LOCATIONS:
Overall Officials: Duane B Corbett, PhD, Study Director — Kent State University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Corbett DB, Fennell C, Peroutky K, Kingsley JD, Glickman EL. The effects of a 12-week worksite physical activity intervention on anthropometric indices, blood pressure indices, and plasma biomarkers of cardiovascular disease risk among university employees. BMC Res Notes. 2018 Jan 29;11(1):80. doi: 10.1186/s13104-018-3151-x. PMID 29378632